CLINICAL TRIAL: NCT04586816
Title: Randomized, Double-Blind Evaluation of Maple Leaf Extract (Maplifa) for Photoaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Verdure Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 005 (Sivamani)
Record Dates: First submitted 2020-05-11; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Photoaging; Hyperpigmentation; Rhytides
Keywords: maple leaf extract; skincare; photoaging; hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Healthy females ages 30-70 with Fitzpatrick skin type I-IV
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vehicle only-placebo (Placebo Comparator): Vehicle cream base containing no maple leaf extract to be applied twice daily to the face
  Interventions: Combination Product: vehicle
- 1% red maple leaf extract (Experimental): lotion preparation with 1% red maple leaf extract to be applied twice daily to the face
  Interventions: Combination Product: 1% red maple leaf extract in cream base
- 5% red maple leaf extract (Experimental): lotion preparation with 5% red maple leaf extract to be applied twice daily to the face
  Interventions: Combination Product: 5% red maple leaf extract

INTERVENTIONS:
Combination Product: 1% red maple leaf extract in cream base — 1% red maple leaf extract is combined in a cream base
  Arms: 1% red maple leaf extract
Combination Product: 5% red maple leaf extract — 5% red maple leaf extract is combined in a cream base
  Arms: 5% red maple leaf extract
Combination Product: vehicle — vehicle cream base only
  Arms: vehicle only-placebo

SUMMARY:
Recent research has reported that the maple leaf extract exhibits anti-aging effects by inhibiting elastase activity, thereby preventing the breakdown of elastin and interfering with the formation of wrinkles. Red maple leaf extract contains phenolic compounds known as glucitol-core-containing gallotannins (GCGs) which help reduce the appearance of wrinkles and may decrease skin inflammation, dark spots and pigmentation. The objective of this study is to examine the effects of topical Maplifa on the cosmetic appearance of facial lines, redness and skin tone.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 30-70
* Individuals with Fitzpatrick skin type I-IV

Exclusion Criteria:

* Individuals who have been on any medication that has caused a change in skin pigmentation based on the opinion of the investigator
* Individuals who have history of acute or chronic disease that would likely interfere with or increase the risk on study participation at the discretion of the investigator
* Individuals who have participated in any other clinical studies using the same test sites (face) and hand in the past 14 days
* Individuals who are pregnant, breast feeding or planning a pregnancy within one month. (There is no concern for risk to fetus but pregnancy can alter skin pigmentation).
* Female volunteers who have started a new hormonal birth control agent or had a change in their hormonal birth control agent within the past 60 days
* Individuals who have had any medical or cosmetic procedure, such as laser resurfacing, or plastic surgery to the test site (face) within the last 6 months. This includes botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
* Individuals who are currently using or during the past 30 days have used a retinoid such as Retin A, or other Rx/OTC Retinyl A or currently using or during the past 14 days have used hydroquinone (skin lightening)
* Individuals with a known history of hypersensitivity to any ingredients to the cosmetic agent that is being assessed
* Individuals who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study at the discretion of the investigator.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Pigmentation on SkinColorCatch | At 4 weeks (end of study)
  Assessment of pigmentation based on melanin measurement on SkinColorCatch (arbitrary units set by technology)
Clinical grading of Hyperpigmentation | At 4 weeks (end of study)
  Assessment of hyperpigmentation based on clinical grading (categories 0-5) by blinded evaluator
Erythema on SkinColorCatch | At 4 weeks (end of study)
  Assessment of erythema based on SkinColorCatch (arbitrary units set by technology)
Clinical grading of Erythema | At 4 weeks (end of study)
  Assessment of erythema based on clinical grading (categories 0-5) by blinded evaluator

SECONDARY OUTCOMES:
Centrofacial redness | At 4 weeks (end of study)
  Image-based analysis of redness [Skinmap level Degree of Intensity (%) on BTBP Clarity Research 3D System]
Appearance of wrinkles | At 4 weeks (end of study)
  Image-based analysis of wrinkles (Average severity - unitless on BTBP Clarity Research 3D System)

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided